CLINICAL TRIAL: NCT01852058
Title: Long-term Extension Study of BOTOX® in the Treatment of Urinary Incontinence Due to Neurogenic Detrusor Overactivity in Patients 5 to 17 Years of Age
Brief Title: A Long-Term Extension Study of OnabotulinumtoxinA (BOTOX®) for Urinary Incontinence Due to Neurogenic Detrusor Overactivity
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 191622-121; 2012-004898-30 (EudraCT Number)
Record Dates: First submitted 2013-05-09; First posted 2013-05-13 (Estimated); Results first posted 2020-05-12 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-04

CONDITIONS: Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- OnabotulinumtoxinA 50 U (Experimental): Following treatment with onabotulinumtoxinA (botulinum toxin Type A) 50 U (not to exceed 6 U/kg) intramuscular injection into the detrusor wall in study 120, participants were eligible for retreatments in this study as needed with a minimum 12-week interval between doses for a maximum of 3 retreatments. Blinded dose increases (one level) were allowed based on clinical response from cycle to cycle (not to exceed 6 U/kg).
  Interventions: Biological: OnabotulinumtoxinA
- OnabotulinumtoxinA 100 U (Experimental): Following treatment with onabotulinumtoxinA (botulinum toxin Type A) 100 U (not to exceed 6 U/kg) intramuscular injection into the detrusor wall in study 120, participants were eligible for retreatments in this study as needed with a minimum 12-week interval between doses for a maximum of 3 retreatments. Blinded dose increases (one level) were allowed based on clinical response from cycle to cycle (not to exceed 6 U/kg).
  Interventions: Biological: OnabotulinumtoxinA
- OnabotulinumtoxinA 200 U (Experimental): Following treatment with onabotulinumtoxinA (botulinum toxin Type A) 200 U (not to exceed 6 U/kg) intramuscular injection into the detrusor wall in study 120, participants were eligible for retreatments in this study as needed with a minimum 12-week interval between doses for a maximum of 3 retreatments. Blinded dose increases (one level) were allowed based on clinical response from cycle to cycle (not to exceed 6 U/kg).
  Interventions: Biological: OnabotulinumtoxinA

INTERVENTIONS:
Biological: OnabotulinumtoxinA — OnabotulinumtoxinA injected into the detrusor wall. Treatments were administered as needed with a minimum of a 12-week interval between doses.
  Other Names: BOTOX®; botulinum toxin Type A

SUMMARY:
This study will evaluate the long-term safety and efficacy of onabotulinumtoxinA (botulinum toxin Type A; BOTOX®) for the treatment of urinary incontinence due to neurogenic detrusor overactivity in participants who successfully completed Study 191622-120 (NCT01852045).

ELIGIBILITY:
Inclusion Criteria:

* Successfully completed participation in Study 191622-120
* Aged ≥ 5 years to ≤ 17 years at the time of entry into Study 191622-120
* Regularly using clean intermittent catheterization to empty the bladder

Exclusion Criteria:

* Myasthenia gravis, Eaton-Lambert syndrome, or amyotrophic lateral sclerosis
* Current or planned use of a baclofen pump
* Current or planned use of an electrostimulation/neuromodulation device for urinary incontinence
* Use of an indwelling catheter for urinary incontinence instead of using clean intermittent catheterization to empty the bladder
* Previous or current use of botulinum toxin therapy of any serotype for any urological condition, or treatment with botulinum toxin of any serotype for any other condition since entering study 191622-120

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 95 (Actual)
Dates: Start 2014-01-11 (Actual); Primary Completion 2018-11-22 (Actual); Study Completion 2019-10-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brenda Jenkins, Study Director — Allergan
Locations (30):
- United States (14):
  - University of Alabama at Birmingham Division of Urology Research Office, Birmingham, Alabama
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - William Beaumont Hospital Research Institute, Royal Oak, Michigan
  - St. Louis Children's Hospital Division of Urology, St Louis, Missouri
  - Pediatric Urology Associates, PC, Tarrytown, New York
  - McKay Urology Carolinas Medical Center, Charlotte, North Carolina
  - Duke University, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center Cincinnati Center for Clinical Research and Outpatient Clinic, Cincinnati, Ohio
  - Oklahoma Children's Hospital, Oklahoma City, Oklahoma
  - Medical University of South Carolina, Charleston, South Carolina
  - Children's Hospital of Wisconsin Department of Pediatric Urology, Milwaukee, Wisconsin
- Belgium (3):
  - UZ Antwerpen, Antwerp
  - Ghent University Hospital, Ghent
  - UZ Leuven, Leuven
- Canada (2):
  - McMaster University Medical Centre, Hamilton, Ontario
  - CHU Sainte Justine, Montreal, Quebec
- Czechia (2):
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Fakultni nemocnice Olomouc, Olomouc
- France (3):
  - Hopital Pellegrin - Enfants, Bordeaux
  - CHU de Limoges - HÃ´pital MÃ¨re et l'Enfant, Limoges
  - Hôpital Necker Enfants-Malades, Paris
- Italy (2):
  - Seconda Università di Napoli, Naples
  - Bambin Gesù- Ospedale Pediatrico, Rome
- Poland (3):
  - Copernicus Podmiot Leczniczy Sp. z o. o. Kliniczny Oddział Chirurgii i Urologii Dzieci i Młodzieży GUMed, Gdansk
  - Specjalistyczny Gabinet Lekarski, Poznan
  - Medical University of Wroclaw, Wroclaw
- University of Ankara, Ankara, Turkey (Türkiye)

REFERENCES:
- See also: More Information — http://www.allerganclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who successfully completed Study 191622-120 (NCT01852045) were enrolled in this study and were followed for up to an additional 60 weeks.
Pre-assignment Details: Data from the participant's participation in this extension Study 191622-121 (121) were integrated with the corresponding participant's data from the preceding Study 191622-120 (120).
Groups:
- OnabotulinumtoxinA 50 U (Treatment Cycle 1): OnabotulinumtoxinA (botulinum toxin Type A) 50 U (not to exceed 6 U/kg) injected into the detrusor wall on Day 1 in Treatment Cycle 1. Participants were eligible for retreatment after Week 12 if qualified. Blinded dose increases (one level) were allowed based on clinical response from cycle to cycle (not to exceed 6 U/kg).
- OnabotulinumtoxinA 100 U (Treatment Cycle 1): OnabotulinumtoxinA (botulinum toxin Type A) 100 U (not to exceed 6 U/kg) injected into the detrusor wall on Day 1 in Treatment Cycle 1. Participants were eligible for retreatment after Week 12 if qualified. Blinded dose increases (one level) were allowed based on clinical response from cycle to cycle (not to exceed 6 U/kg).
- OnabotulinumtoxinA 200 U (Treatment Cycle 1): OnabotulinumtoxinA (botulinum toxin Type A) 200 U (not to exceed 6 U/kg) injected into the detrusor wall on Day 1 in Treatment Cycle 1. Participants were eligible for retreatment after Week 12 if qualified. Blinded dose increases (one level) were allowed based on clinical response from cycle to cycle (not to exceed 6 U/kg).
- OnabotulinumtoxinA 50 U (Treatment Cycle 2): OnabotulinumtoxinA (botulinum toxin Type A) 50 U (not to exceed 6 U/kg) injected into the detrusor wall on Day 1 in Treatment Cycle 2. Participants were eligible for retreatment after Week 12 if qualified. Blinded dose increases (one level) were allowed based on clinical response from cycle to cycle (not to exceed 6 U/kg).
- OnabotulinumtoxinA 100 U (Treatment Cycle 2): OnabotulinumtoxinA (botulinum toxin Type A) 100 U (not to exceed 6 U/kg) injected into the detrusor wall on Day 1 in Treatment Cycle 2. Participants were eligible for retreatment after Week 12 if qualified. Blinded dose increases (one level) were allowed based on clinical response from cycle to cycle (not to exceed 6 U/kg).
- OnabotulinumtoxinA 200 U (Treatment Cycle 2): OnabotulinumtoxinA (botulinum toxin Type A) 200 U (not to exceed 6 U/kg) injected into the detrusor wall on Day 1 in Treatment Cycle 2. Participants were eligible for retreatment after Week 12 if qualified. Blinded dose increases (one level) were allowed based on clinical response from cycle to cycle (not to exceed 6 U/kg).
- OnabotulinumtoxinA 50 U (Treatment Cycle 3): OnabotulinumtoxinA (botulinum toxin Type A) 50 U (not to exceed 6 U/kg) injected into the detrusor wall on Day 1 in Treatment Cycle 3. Participants were eligible for retreatment after Week 12 if qualified. Blinded dose increases (one level) were allowed based on clinical response from cycle to cycle (not to exceed 6 U/kg).
- OnabotulinumtoxinA 100 U (Treatment Cycle 3): OnabotulinumtoxinA (botulinum toxin Type A) 100 U (not to exceed 6 U/kg) injected into the detrusor wall on Day 1 in Treatment Cycle 3. Participants were eligible for retreatment after Week 12 if qualified. Blinded dose increases (one level) were allowed based on clinical response from cycle to cycle (not to exceed 6 U/kg).
- OnabotulinumtoxinA 200 U (Treatment Cycle 3): OnabotulinumtoxinA (botulinum toxin Type A) 200 U (not to exceed 6 U/kg) injected into the detrusor wall on Day 1 in Treatment Cycle 3. Participants were eligible for retreatment after Week 12 if qualified. Blinded dose increases (one level) were allowed based on clinical response from cycle to cycle (not to exceed 6 U/kg).
- OnabotulinumtoxinA 50 U (Treatment Cycle 4): OnabotulinumtoxinA (botulinum toxin Type A) 50 U (not to exceed 6 U/kg) injected into the detrusor wall on Day 1 in Treatment Cycle 4. Blinded dose increases (one level) were allowed based on clinical response from cycle to cycle (not to exceed 6 U/kg).
- OnabotulinumtoxinA 100 U (Treatment Cycle 4): OnabotulinumtoxinA (botulinum toxin Type A) 100 U (not to exceed 6 U/kg) injected into the detrusor wall on Day 1 in Treatment Cycle 4. Blinded dose increases (one level) were allowed based on clinical response from cycle to cycle (not to exceed 6 U/kg).
- OnabotulinumtoxinA 200 U (Treatment Cycle 4): OnabotulinumtoxinA (botulinum toxin Type A) 200 U (not to exceed 6 U/kg) injected into the detrusor wall on Day 1 in Treatment Cycle 4. Blinded dose increases (one level) were allowed based on clinical response from cycle to cycle (not to exceed 6 U/kg).
Period: Treatment Cycle 1, Occurred in Study 120
Arm/Group | OnabotulinumtoxinA 50 U (Treatment Cycle 1) | OnabotulinumtoxinA 100 U (Treatment Cycle 1) | OnabotulinumtoxinA 200 U (Treatment Cycle 1) | OnabotulinumtoxinA 50 U (Treatment Cycle 2) | OnabotulinumtoxinA 100 U (Treatment Cycle 2) | OnabotulinumtoxinA 200 U (Treatment Cycle 2) | OnabotulinumtoxinA 50 U (Treatment Cycle 3) | OnabotulinumtoxinA 100 U (Treatment Cycle 3) | OnabotulinumtoxinA 200 U (Treatment Cycle 3) | OnabotulinumtoxinA 50 U (Treatment Cycle 4) | OnabotulinumtoxinA 100 U (Treatment Cycle 4) | OnabotulinumtoxinA 200 U (Treatment Cycle 4)
Started | 31 | 39 | 25 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed (Completed=Completed the entire study in this Cycle) | 30 | 39 | 25 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Cycle2:Retreatment 1,Study 121
Arm/Group | OnabotulinumtoxinA 50 U (Treatment Cycle 1) | OnabotulinumtoxinA 100 U (Treatment Cycle 1) | OnabotulinumtoxinA 200 U (Treatment Cycle 1) | OnabotulinumtoxinA 50 U (Treatment Cycle 2) | OnabotulinumtoxinA 100 U (Treatment Cycle 2) | OnabotulinumtoxinA 200 U (Treatment Cycle 2) | OnabotulinumtoxinA 50 U (Treatment Cycle 3) | OnabotulinumtoxinA 100 U (Treatment Cycle 3) | OnabotulinumtoxinA 200 U (Treatment Cycle 3) | OnabotulinumtoxinA 50 U (Treatment Cycle 4) | OnabotulinumtoxinA 100 U (Treatment Cycle 4) | OnabotulinumtoxinA 200 U (Treatment Cycle 4)
Started | 0 | 0 | 0 | 9 | 45 | 36 | 0 | 0 | 0 | 0 | 0 | 0
Completed (Completed=Completed the entire study in this Cycle) | 0 | 0 | 0 | 8 | 38 | 27 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 1 | 7 | 9 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Deviation | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Reason not Specified | 0 | 0 | 0 | 0 | 1 | 7 | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Cycle3:Retreatment 2,Study 121
Arm/Group | OnabotulinumtoxinA 50 U (Treatment Cycle 1) | OnabotulinumtoxinA 100 U (Treatment Cycle 1) | OnabotulinumtoxinA 200 U (Treatment Cycle 1) | OnabotulinumtoxinA 50 U (Treatment Cycle 2) | OnabotulinumtoxinA 100 U (Treatment Cycle 2) | OnabotulinumtoxinA 200 U (Treatment Cycle 2) | OnabotulinumtoxinA 50 U (Treatment Cycle 3) | OnabotulinumtoxinA 100 U (Treatment Cycle 3) | OnabotulinumtoxinA 200 U (Treatment Cycle 3) | OnabotulinumtoxinA 50 U (Treatment Cycle 4) | OnabotulinumtoxinA 100 U (Treatment Cycle 4) | OnabotulinumtoxinA 200 U (Treatment Cycle 4)
Started | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 16 | 34 | 0 | 0 | 0
Completed (Completed=Completed the entire study in this Cycle) | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 15 | 33 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Reason Not Specified | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Period: Treatment Cycle4:Retreatment 3,Study 121
Arm/Group | OnabotulinumtoxinA 50 U (Treatment Cycle 1) | OnabotulinumtoxinA 100 U (Treatment Cycle 1) | OnabotulinumtoxinA 200 U (Treatment Cycle 1) | OnabotulinumtoxinA 50 U (Treatment Cycle 2) | OnabotulinumtoxinA 100 U (Treatment Cycle 2) | OnabotulinumtoxinA 200 U (Treatment Cycle 2) | OnabotulinumtoxinA 50 U (Treatment Cycle 3) | OnabotulinumtoxinA 100 U (Treatment Cycle 3) | OnabotulinumtoxinA 200 U (Treatment Cycle 3) | OnabotulinumtoxinA 50 U (Treatment Cycle 4) | OnabotulinumtoxinA 100 U (Treatment Cycle 4) | OnabotulinumtoxinA 200 U (Treatment Cycle 4)
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 4 | 4
Completed (Completed=Completed the entire study in this Cycle) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: BOTOX-treated Population included all participants enrolled into the extension study who received at least 1 BOTOX treatment over the course of the total evaluation period, starting from their first treatment in Study 120.
Groups:
- Total: Total of all reporting groups
Arm/Group | OnabotulinumtoxinA 50 U | OnabotulinumtoxinA 100 U | OnabotulinumtoxinA 200 U | Total
Number analyzed (Participants) | 31 | 39 | 25 | 95
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.7 (3.49) | 10.8 (3.36) | 11.7 (3.22) | 11.3 (3.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 14 | 13 | 44
  Male | 14 | 25 | 12 | 51
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 22 | 28 | 18 | 68
  Black or African American | 6 | 3 | 2 | 11
  Asian | 1 | 2 | 0 | 3
  Hispanic | 1 | 3 | 3 | 7
  Other | 1 | 3 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Change From Study Baseline in the Daily Normalized Daytime Average Number of Urinary Incontinence Episodes in Treatment Cycle 1
Description: Urinary incontinence was defined as involuntary loss of urine as recorded by the participant in a bladder diary during 2 consecutive days in the week prior to the study visit (normalized to a 12 hour daytime period). Daytime is defined as the time between waking up to start the day and going to bed to sleep for the night. The number of daily daytime incontinence episodes were averaged during the 2-day period. A negative change from Baseline indicates improvement. Data are summarized under the respective treatments that participants received in the corresponding treatment cycle.
Time Frame: Study Baseline (Prior to Day 1 in Study 120) to 2 consecutive days in the week prior to Week 6 in Treatment Cycle 1
Population: BOTOX-treated Population included all participants enrolled into the extension study who received at least 1 BOTOX treatment over the course of the total evaluation period, starting from their first treatment in Study 120. Number analyzed is the number of participants with evaluable data at the given timepoint.
Measure: Mean (Standard Deviation); unit: urinary incontinence episodes per day
Arm/Group | OnabotulinumtoxinA 50 U (Treatment Cycle 1) | OnabotulinumtoxinA 100 U (Treatment Cycle 1) | OnabotulinumtoxinA 200 U (Treatment Cycle 1)
Number analyzed (Participants) | 31 | 39 | 25
urinary incontinence episodes per day
  Baseline | 2.66 (0.876) | 2.97 (1.135) | 3.99 (5.492)
  Change from Baseline to Week 6: number analyzed (Participants) | 30 | 36 | 23
  Change from Baseline to Week 6 | -1.19 (1.156) | -1.39 (1.585) | -2.19 (5.738)

2. Primary Outcome: Change From Study Baseline in the Daily Normalized Daytime Average Number of Urinary Incontinence Episodes in Treatment Cycle 2
Description: as for outcome 1
Time Frame: Study Baseline (Prior to Day 1 in Study 120) to 2 consecutive days in the week prior to Week 6 in Treatment Cycle 2
Population: BOTOX-treated Population included all participants enrolled into the extension study who received at least 1 BOTOX treatment over the course of the total evaluation period, starting from their first treatment in Study 120. Number analyzed is the number of participants with evaluable data at the given time point.
Measure: Mean (Standard Deviation); unit: urinary incontinence episodes per day
Arm/Group | OnabotulinumtoxinA 50 U (Treatment Cycle 2) | OnabotulinumtoxinA 100 U (Treatment Cycle 2) | OnabotulinumtoxinA 200 U (Treatment Cycle 2)
Number analyzed (Participants) | 9 | 45 | 36
urinary incontinence episodes per day
  Baseline | 2.57 (0.937) | 2.80 (0.915) | 3.83 (4.623)
  Change from Baseline to Week 6: number analyzed (Participants) | 6 | 44 | 34
  Change from Baseline to Week 6 | -1.07 (2.092) | -1.70 (1.331) | -1.64 (1.906)

3. Primary Outcome: Change From Study Baseline in the Daily Normalized Daytime Average Number of Urinary Incontinence Episodes in Treatment Cycle 3
Description: as for outcome 1
Time Frame: Study Baseline (Prior to Day 1 in Study 120) to 2 consecutive days in the week prior to Week 6 in Treatment Cycle 3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: urinary incontinence episodes per day
Arm/Group | OnabotulinumtoxinA 50 U (Treatment Cycle 3) | OnabotulinumtoxinA 100 U (Treatment Cycle 3) | OnabotulinumtoxinA 200 U (Treatment Cycle 3)
Number analyzed (Participants) | 5 | 16 | 34
urinary incontinence episodes per day
  Baseline | 2.48 (0.228) | 2.94 (0.923) | 3.80 (4.678)
  Change from Baseline to Week 6: number analyzed (Participants) | 5 | 16 | 33
  Change from Baseline to Week 6 | -1.92 (0.858) | -1.73 (1.057) | -2.74 (4.833)

4. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious Treatment Emergent Adverse Events (STEAEs)
Description: An adverse event is any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with use of a medicinal (investigational) product, whether or not related to medicinal (investigational) product. A serious adverse event (SAE) is any AE that resulted in death, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, life threatening, a congenital anomaly/birth defect, or an important medical event. A TEAE or STEAE is defined as any new AE or worsening of an existing condition after initiation of treatment. Data are summarized under the respective treatments that participants received in the corresponding treatment cycles.
Time Frame: First injection on Day 1 in Study 120 through completion of Study 121 (Up to 108 weeks)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | OnabotulinumtoxinA 50 U (Treatment Cycle 1) | OnabotulinumtoxinA 100 U (Treatment Cycle 1) | OnabotulinumtoxinA 200 U (Treatment Cycle 1) | OnabotulinumtoxinA 50 U (Treatment Cycle 2) | OnabotulinumtoxinA 100 U (Treatment Cycle 2) | OnabotulinumtoxinA 200 U (Treatment Cycle 2) | OnabotulinumtoxinA 50 U (Treatment Cycle 3) | OnabotulinumtoxinA 100 U (Treatment Cycle 3) | OnabotulinumtoxinA 200 U (Treatment Cycle 3) | OnabotulinumtoxinA 50 U (Treatment Cycle 4) | OnabotulinumtoxinA 100 U (Treatment Cycle 4) | OnabotulinumtoxinA 200 U (Treatment Cycle 4)
Number analyzed (Participants) | 31 | 39 | 25 | 9 | 45 | 36 | 5 | 16 | 34 | 3 | 4 | 4
Participants
  TEAEs | 23 | 31 | 19 | 7 | 34 | 31 | 4 | 10 | 21 | 3 | 2 | 4
  STEAEs | 2 | 3 | 1 | 0 | 5 | 6 | 0 | 1 | 2 | 0 | 0 | 0

5. Secondary Outcome: Percentage of Participants With ≥ 50%, ≥ 75%, ≥ 90%, and ≥ 100% Reduction From Baseline in the Number of Normalized Daytime Urinary Incontinence Episodes in Treatment Cycle 1
Description: Urinary incontinence was defined as involuntary loss of urine as recorded by the participant in a bladder diary during 2 consecutive days in the week prior to the study visit (normalized to a 12 hour daytime period). Daytime is defined as the time between waking up to start the day and going to bed to sleep for the night. The number of daily incontinence episodes were averaged during the 2-day period. Data are summarized under the respective treatments that participants received in the corresponding treatment cycle.
Time Frame: Study Baseline (Prior to Day 1 in Study 120) to 2 consecutive days in the week prior to Week 6 in Treatment Cycle 1
Population: BOTOX-treated Population included all participants enrolled into extension study who received at least 1 BOTOX treatment over the course of total evaluation period, starting from their first treatment in Study 120. Number analyzed is the number of participants with evaluable data for the specific category.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | OnabotulinumtoxinA 50 U (Treatment Cycle 1) | OnabotulinumtoxinA 100 U (Treatment Cycle 1) | OnabotulinumtoxinA 200 U (Treatment Cycle 1)
Number analyzed (Participants) | 31 | 39 | 25
percentage of participants
  ≥50% Reduction from Baseline to Week 6: number analyzed (Participants) | 30 | 36 | 23
  ≥50% Reduction from Baseline to Week 6 | 53.3 [34.33 to 71.66] | 55.6 [38.10 to 72.06] | 52.2 [30.59 to 73.18]
  ≥75% Reduction from Baseline to Week 6: number analyzed (Participants) | 30 | 36 | 23
  ≥75% Reduction from Baseline to Week 6 | 30.0 [14.73 to 49.40] | 41.7 [25.51 to 59.24] | 39.1 [19.71 to 61.46]
  ≥90% Reduction from Baseline to Week 6: number analyzed (Participants) | 30 | 36 | 23
  ≥90% Reduction from Baseline to Week 6 | 26.7 [12.28 to 45.89] | 30.6 [16.35 to 48.11] | 30.4 [13.21 to 52.92]
  ≥100% Reduction from Baseline to Week 6: number analyzed (Participants) | 30 | 36 | 23
  ≥100% Reduction from Baseline to Week 6 | 26.7 [12.28 to 45.89] | 27.8 [14.20 to 45.19] | 26.1 [10.23 to 48.41]

6. Secondary Outcome: Percentage of Participants With ≥ 50%, ≥ 75%, ≥ 90%, and ≥ 100% Reduction From Baseline in the Number of Normalized Daytime Urinary Incontinence Episodes in Treatment Cycle 2
Description: as for outcome 5
Time Frame: Study Baseline (Prior to Day 1 in Study 120) to 2 consecutive days in the week prior to Week 6 in Treatment Cycle 2
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | OnabotulinumtoxinA 50 U (Treatment Cycle 2) | OnabotulinumtoxinA 100 U (Treatment Cycle 2) | OnabotulinumtoxinA 200 U (Treatment Cycle 2)
Number analyzed (Participants) | 9 | 45 | 36
percentage of participants
  ≥50% Reduction from Baseline to Week 6: number analyzed (Participants) | 6 | 44 | 34
  ≥50% Reduction from Baseline to Week 6 | 66.7 [22.28 to 95.67] | 65.9 [50.08 to 79.51] | 58.8 [40.70 to 75.35]
  ≥75% Reduction from Baseline to Week 6: number analyzed (Participants) | 6 | 44 | 34
  ≥75% Reduction from Baseline to Week 6 | 50.0 [11.81 to 88.19] | 43.2 [28.35 to 58.97] | 47.1 [29.78 to 64.87]
  ≥90% Reduction from Baseline to Week 6: number analyzed (Participants) | 6 | 44 | 34
  ≥90% Reduction from Baseline to Week 6 | 50.0 [11.81 to 88.19] | 27.3 [14.96 to 42.79] | 41.2 [24.65 to 59.30]
  ≥100% Reduction from Baseline to Week 6: number analyzed (Participants) | 6 | 44 | 34
  ≥100% Reduction from Baseline to Week 6 | 50.0 [11.81 to 88.19] | 25.0 [13.19 to 40.34] | 38.2 [22.17 to 56.44]

7. Secondary Outcome: Percentage of Participants With ≥ 50%, ≥ 75%, ≥ 90%, and ≥ 100% Reduction From Baseline in the Number of Normalized Daytime Urinary Incontinence Episodes in Treatment Cycle 3
Description: as for outcome 5
Time Frame: Study Baseline (Prior to Day 1 in Study 120) to 2 consecutive days in the week prior to Week 6 in Treatment Cycle 3
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | OnabotulinumtoxinA 50 U (Treatment Cycle 3) | OnabotulinumtoxinA 100 U (Treatment Cycle 3) | OnabotulinumtoxinA 200 U (Treatment Cycle 3)
Number analyzed (Participants) | 5 | 16 | 34
percentage of participants
  ≥50% Reduction from Baseline at Week 6: number analyzed (Participants) | 5 | 16 | 33
  ≥50% Reduction from Baseline at Week 6 | 60.0 [14.66 to 94.73] | 75.0 [47.62 to 92.73] | 69.7 [51.29 to 84.41]
  ≥75% Reduction from Baseline at Week 6: number analyzed (Participants) | 5 | 16 | 33
  ≥75% Reduction from Baseline at Week 6 | 60.0 [14.66 to 94.73] | 37.5 [15.20 to 64.57] | 39.4 [22.91 to 57.86]
  ≥90% Reduction from Baseline at Week 6: number analyzed (Participants) | 5 | 16 | 33
  ≥90% Reduction from Baseline at Week 6 | 60.0 [14.66 to 94.73] | 18.8 [4.05 to 45.65] | 33.3 [17.96 to 51.83]
  ≥100% Reduction from Baseline at Week 6: number analyzed (Participants) | 5 | 16 | 33
  ≥100% Reduction from Baseline at Week 6 | 60.0 [14.66 to 94.73] | 18.8 [4.05 to 45.65] | 30.3 [15.59 to 48.71]

8. Secondary Outcome: Change From Baseline in Average Urine Volume at First Morning Catheterization in Treatment Cycle 1
Description: The change in urine volume at first morning catherization was recorded by the participant in a bladder diary in the 2 consecutive days during the week prior to the study visit. The daily values were averaged during the 2-day period. A positive change from Baseline indicates improvement. Data are summarized under the respective treatments that participants received in the corresponding treatment cycle.
Time Frame: Baseline (Prior to Day 1 in Study 120) to 2 consecutive days in the week prior to Week 6 in Treatment Cycle 1
Population: BOTOX-treated Population included all participants enrolled into extension study who received >=1 BOTOX treatment over course of total evaluation period, starting from their first treatment in Study 120. Overall number of participants analyzed is the number of participants with data available for analyses.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | OnabotulinumtoxinA 50 U (Treatment Cycle 1) | OnabotulinumtoxinA 100 U (Treatment Cycle 1) | OnabotulinumtoxinA 200 U (Treatment Cycle 1)
Number analyzed (Participants) | 30 | 36 | 21
mL | 14.68 (88.146) | 39.88 (72.787) | 96.90 (120.429)

9. Secondary Outcome: Change From Baseline in Average Urine Volume at First Morning Catheterization in Treatment Cycle 2
Description: as for outcome 8
Time Frame: Baseline (Prior to Day 1 in Study 120) to 2 consecutive days in the week prior to Week 6 in Treatment Cycle 2
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | OnabotulinumtoxinA 50 U (Treatment Cycle 2) | OnabotulinumtoxinA 100 U (Treatment Cycle 2) | OnabotulinumtoxinA 200 U (Treatment Cycle 2)
Number analyzed (Participants) | 6 | 43 | 31
mL | 7.92 (148.597) | 79.53 (106.794) | 35.34 (98.209)

10. Secondary Outcome: Change From Baseline in Average Urine Volume at First Morning Catheterization in Treatment Cycle 3
Description: as for outcome 8
Time Frame: Baseline (Prior to Day 1 in Study 120) to 2 consecutive days in the week prior to Week 6 in Treatment Cycle 3
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | OnabotulinumtoxinA 50 U (Treatment Cycle 3) | OnabotulinumtoxinA 100 U (Treatment Cycle 3) | OnabotulinumtoxinA 200 U (Treatment Cycle 3)
Number analyzed (Participants) | 5 | 10 | 31
mL | 58.50 (22.749) | 57.86 (74.762) | 92.39 (147.322)

11. Secondary Outcome: Percentage of Participants With Night Time Urinary Incontinence in Treatment Cycle 1
Description: Urinary incontinence was defined as involuntary loss of urine. Night time urinary incontinence was recorded by the participant on the bladder diary as a presence or absence of urinary leakage upon waking, for 2 consecutive days in the week prior to the week 6 visit. Night time was defined as the time between going to bed to sleep for the night and waking up to start the day. The percentage of participants with night time urinary incontinence is presented in categories 0, 1, and 2 nights. Data are summarized under the respective treatments that participants received in the corresponding treatment cycle.
Time Frame: Baseline (Prior to Day 1 in Study 120) and 2 consecutive days in the week prior to Week 6 in Treatment Cycle 1
Population: BOTOX-treated Population included all participants enrolled into extension study who received >= 1 BOTOX treatment over course of total evaluation period, starting from their first treatment in Study 120. Number analyzed is the number of participants with data available for analyses at the given time point.
Measure: Number; unit: percentage of participants
Arm/Group | OnabotulinumtoxinA 50 U (Treatment Cycle 1) | OnabotulinumtoxinA 100 U (Treatment Cycle 1) | OnabotulinumtoxinA 200 U (Treatment Cycle 1)
Number analyzed (Participants) | 31 | 39 | 25
percentage of participants
  0 Nights of Incontinence at Baseline: number analyzed (Participants) | 31 | 39 | 23
  0 Nights of Incontinence at Baseline | 0.0 | 15.4 | 4.3
  0 Nights of Incontinence at Week 6: number analyzed (Participants) | 30 | 37 | 24
  0 Nights of Incontinence at Week 6 | 30.0 | 37.8 | 25.0
  1 Night of Incontinence at Baseline: number analyzed (Participants) | 31 | 39 | 23
  1 Night of Incontinence at Baseline | 12.9 | 2.6 | 17.4
  1 Night of Incontinence at Week 6: number analyzed (Participants) | 30 | 37 | 24
  1 Night of Incontinence at Week 6 | 20.0 | 16.2 | 29.2
  2 Nights of Incontinence at Baseline: number analyzed (Participants) | 31 | 39 | 23
  2 Nights of Incontinence at Baseline | 87.1 | 82.1 | 78.3
  2 Nights of Incontinence at Week 6: number analyzed (Participants) | 30 | 37 | 24
  2 Nights of Incontinence at Week 6 | 50.0 | 45.9 | 45.8

12. Secondary Outcome: Percentage of Participants With Night Time Urinary Incontinence in Treatment Cycle 2
Description: as for outcome 11
Time Frame: Baseline (Prior to Day 1 in Study 120) and 2 consecutive days in the week prior to Week 6 in Treatment Cycle 2
Population: as for outcome 11
Measure: Number; unit: percentage of participants
Arm/Group | OnabotulinumtoxinA 50 U (Treatment Cycle 2) | OnabotulinumtoxinA 100 U (Treatment Cycle 2) | OnabotulinumtoxinA 200 U (Treatment Cycle 2)
Number analyzed (Participants) | 9 | 45 | 36
percentage of participants
  0 Nights of Incontinence at Baseline: number analyzed (Participants) | 9 | 45 | 34
  0 Nights of Incontinence at Baseline | 0.0 | 8.9 | 5.9
  0 Nights of Incontinence at Week 6: number analyzed (Participants) | 6 | 44 | 34
  0 Nights of Incontinence at Week 6 | 66.7 | 34.1 | 23.5
  1 Night of Incontinence at Baseline: number analyzed (Participants) | 9 | 45 | 34
  1 Night of Incontinence at Baseline | 22.2 | 6.7 | 8.8
  1 Night of Incontinence at Week 6: number analyzed (Participants) | 6 | 44 | 34
  1 Night of Incontinence at Week 6 | 16.7 | 22.7 | 8.8
  2 Nights of Incontinence at Baseline: number analyzed (Participants) | 9 | 45 | 34
  2 Nights of Incontinence at Baseline | 77.8 | 84.4 | 85.3
  2 Nights of Incontinence at Week 6: number analyzed (Participants) | 6 | 44 | 34
  2 Nights of Incontinence at Week 6 | 16.7 | 43.2 | 67.6

13. Secondary Outcome: Percentage of Participants With Night Time Urinary Incontinence in Treatment Cycle 3
Description: as for outcome 11
Time Frame: Baseline (Prior to Day 1 in Study 120) and 2 consecutive days in the week prior to Week 6 in Treatment Cycle 3
Population: as for outcome 11
Measure: Number; unit: percentage of participants
Arm/Group | OnabotulinumtoxinA 50 U (Treatment Cycle 3) | OnabotulinumtoxinA 100 U (Treatment Cycle 3) | OnabotulinumtoxinA 200 U (Treatment Cycle 3)
Number analyzed (Participants) | 5 | 16 | 34
percentage of participants
  0 Nights of Incontinence at Baseline | 0.0 | 12.5 | 5.9
  0 Nights of Incontinence at Week 6: number analyzed (Participants) | 5 | 16 | 33
  0 Nights of Incontinence at Week 6 | 20.0 | 31.3 | 21.2
  1 Night of Incontinence at Baseline | 0.0 | 0.0 | 5.9
  1 Night of Incontinence at Week 6: number analyzed (Participants) | 5 | 16 | 33
  1 Night of Incontinence at Week 6 | 40.0 | 12.5 | 27.3
  2 Nights of Incontinence at Baseline | 100.0 | 87.5 | 88.2
  2 Nights of Incontinence at Week 6: number analyzed (Participants) | 5 | 16 | 33
  2 Nights of Incontinence at Week 6 | 40.0 | 56.3 | 51.5

14. Secondary Outcome: Average Time to Participant's Request for Retreatment
Description: Time to request for re-treatment is the time in weeks between last injection and request for next injection, regardless of fulfillment of the re-treatment criteria. Data are summarized under the respective treatments that participants received across entire study. Data is reported for only participants that had at least one request for retreatment while on a specified BOTOX dose.
Time Frame: First injection on Day 1 in Study 120 through to the date of completion of Study 121 (Up to 108 weeks)
Population: as for outcome 8
Measure: Median (Full Range); unit: weeks
Arm/Group | OnabotulinumtoxinA 50 U | OnabotulinumtoxinA 100 U | OnabotulinumtoxinA 200 U
Number analyzed (Participants) | 30 | 53 | 35
weeks | 24.55 [11.9 to 89.7] | 24.64 [11.7 to 73.3] | 25.43 [11.1 to 78.9]

15. Secondary Outcome: Average Time to Participant's Qualification for Retreatment
Description: The criteria for qualification of retreatment included 1) Participant/parent/caregiver requests retreatment; 2) Participant has a total of at least 2 daytime urinary incontinence episodes over the 2-day bladder diary collection period; 3) At least 12 weeks has elapsed since treatment 1 and 4) Participant has not experienced a serious treatment-related adverse event at any time. Data are summarized under the respective treatments that participants received across entire study. Data is reported for only participants that had at least one request for retreatment while on a specified BOTOX dose.
Time Frame: First injection on Day 1 in Study 120 through to the date of completion of Study 121 (Up to 108 weeks)
Population: as for outcome 8
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | OnabotulinumtoxinA 50 U | OnabotulinumtoxinA 100 U | OnabotulinumtoxinA 200 U
Number analyzed (Participants) | 29 | 53 | 25
weeks | 25.38 [11.9 to 84.4] | 25.43 [11.7 to 76.1] | 26.29 [11.1 to 78.9]

16. Secondary Outcome: Percentage of Participants With Positive Response on Modified Treatment Benefit Scale (TBS) in Treatment Cycle 1
Description: The Modified TBS is a single-item scale which assesses the participant's condition (urinary problems, urinary incontinence) on a 4-point scale where 1 = greatly improved; 2 = improved; 3 = not changed; and 4 = worsened. A participant was considered to have a positive treatment response if they responded to the TBS question as either "greatly improved" or "improved". Data are summarized under the respective treatments that participants received in the corresponding treatment cycle.
Time Frame: Week 6 in Treatment Cycle 1
Population: BOTOX-treated Population included all participants enrolled into extension study who received >=1 BOTOX treatment over course of total evaluation period,starting from their first treatment in Study 120. Overall number of participants analyzed is number of participants with data available for analyses.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | OnabotulinumtoxinA 50 U (Treatment Cycle 1) | OnabotulinumtoxinA 100 U (Treatment Cycle 1) | OnabotulinumtoxinA 200 U (Treatment Cycle 1)
Number analyzed (Participants) | 30 | 35 | 24
percentage of participants | 80.0 [61.43 to 92.29] | 80.0 [63.06 to 91.56] | 75.0 [53.29 to 90.23]

17. Secondary Outcome: Percentage of Participants With Positive Response on Modified Treatment Benefit Scale (TBS) in Treatment Cycle 2
Description: as for outcome 16
Time Frame: Week 6 in Treatment Cycle 2
Population: BOTOX-treated Population included all participants enrolled into extension study who received >=1 BOTOX treatment over course of total evaluation period,starting from their first treatment in Study 120. Overall number of participants analyzed is the number of participants with data available for analyses.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | OnabotulinumtoxinA 50 U (Treatment Cycle 2) | OnabotulinumtoxinA 100 U (Treatment Cycle 2) | OnabotulinumtoxinA 200 U (Treatment Cycle 2)
Number analyzed (Participants) | 8 | 42 | 30
percentage of participants | 75.0 [34.91 to 96.81] | 97.6 [87.43 to 99.94] | 83.3 [65.28 to 94.36]

18. Secondary Outcome: Percentage of Participants With Positive Response on Modified Treatment Benefit Scale (TBS) in Treatment Cycle 3
Description: as for outcome 16
Time Frame: Week 6 in Treatment Cycle 3
Population: as for outcome 17
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | OnabotulinumtoxinA 50 U (Treatment Cycle 3) | OnabotulinumtoxinA 100 U (Treatment Cycle 3) | OnabotulinumtoxinA 200 U (Treatment Cycle 3)
Number analyzed (Participants) | 5 | 15 | 33
percentage of participants | 100 [47.82 to 100.00] | 80.0 [51.91 to 95.67] | 84.8 [68.10 to 94.89]

ADVERSE EVENTS:
Time Frame: First injection on Day 1 in Study 120 through the completion of Study 121 (Up to 108 Weeks)
Description: BOTOX-treated Population included all participants enrolled into the extension study who received at least 1 BOTOX treatment over the course of the total evaluation period, starting from their first treatment in Study 191622-120. Data are summarized under the respective treatments that participants received in the corresponding treatment cycles.
Arm/Group | OnabotulinumtoxinA 50 U (Treatment Cycle 1) | OnabotulinumtoxinA 100 U (Treatment Cycle 1) | OnabotulinumtoxinA 200 U (Treatment Cycle 1) | OnabotulinumtoxinA 50 U (Treatment Cycle 2) | OnabotulinumtoxinA 100 U (Treatment Cycle 2) | OnabotulinumtoxinA 200 U (Treatment Cycle 2) | OnabotulinumtoxinA 50 U (Treatment Cycle 3) | OnabotulinumtoxinA 100 U (Treatment Cycle 3) | OnabotulinumtoxinA 200 U (Treatment Cycle 3) | OnabotulinumtoxinA 50 U (Treatment Cycle 4) | OnabotulinumtoxinA 100 U (Treatment Cycle 4) | OnabotulinumtoxinA 200 U (Treatment Cycle 4)
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/39 | 0/25 | 0/9 | 0/45 | 0/36 | 0/5 | 0/16 | 0/34 | 0/3 | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 2/31 | 3/39 | 1/25 | 0/9 | 5/45 | 6/36 | 0/5 | 1/16 | 2/34 | 0/3 | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 21/31 | 31/39 | 16/25 | 7/9 | 32/45 | 27/36 | 4/5 | 10/16 | 19/34 | 3/3 | 2/4 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OnabotulinumtoxinA 50 U (Treatment Cycle 1) (N=31) | OnabotulinumtoxinA 100 U (Treatment Cycle 1) (N=39) | OnabotulinumtoxinA 200 U (Treatment Cycle 1) (N=25) | OnabotulinumtoxinA 50 U (Treatment Cycle 2) (N=9) | OnabotulinumtoxinA 100 U (Treatment Cycle 2) (N=45) | OnabotulinumtoxinA 200 U (Treatment Cycle 2) (N=36) | OnabotulinumtoxinA 50 U (Treatment Cycle 3) (N=5) | OnabotulinumtoxinA 100 U (Treatment Cycle 3) (N=16) | OnabotulinumtoxinA 200 U (Treatment Cycle 3) (N=34) | OnabotulinumtoxinA 50 U (Treatment Cycle 4) (N=3) | OnabotulinumtoxinA 100 U (Treatment Cycle 4) (N=4) | OnabotulinumtoxinA 200 U (Treatment Cycle 4) (N=4)
Urinary tract infection (Infections and infestations) | 1 | 2 | 0 | 0 | 1 | 2 | 0 | 0 | 2 | 0 | 0 | 0
Encephalitis viral (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hydrocephalus (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bacterial diarrhoea (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Febrile infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fistula (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hip deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Device malfunction (Product Issues) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Epilepsy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | OnabotulinumtoxinA 50 U (Treatment Cycle 1) (N=31) | OnabotulinumtoxinA 100 U (Treatment Cycle 1) (N=39) | OnabotulinumtoxinA 200 U (Treatment Cycle 1) (N=25) | OnabotulinumtoxinA 50 U (Treatment Cycle 2) (N=9) | OnabotulinumtoxinA 100 U (Treatment Cycle 2) (N=45) | OnabotulinumtoxinA 200 U (Treatment Cycle 2) (N=36) | OnabotulinumtoxinA 50 U (Treatment Cycle 3) (N=5) | OnabotulinumtoxinA 100 U (Treatment Cycle 3) (N=16) | OnabotulinumtoxinA 200 U (Treatment Cycle 3) (N=34) | OnabotulinumtoxinA 50 U (Treatment Cycle 4) (N=3) | OnabotulinumtoxinA 100 U (Treatment Cycle 4) (N=4) | OnabotulinumtoxinA 200 U (Treatment Cycle 4) (N=4)
Diarrhoea (Gastrointestinal disorders) | 2 | 2 | 2 | 1 | 2 | 3 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 1 | 1 | 1 | 3 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 2 | 0 | 2 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 5 | 0 | 0 | 6 | 3 | 0 | 0 | 3 | 0 | 1 | 1
Suprapubic pain (General disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 9 | 13 | 5 | 1 | 22 | 6 | 0 | 4 | 6 | 1 | 1 | 0
Bacteriuria (Infections and infestations) | 5 | 7 | 5 | 1 | 9 | 2 | 0 | 3 | 4 | 2 | 0 | 0
Pharyngitis (Infections and infestations) | 3 | 4 | 0 | 0 | 3 | 2 | 0 | 1 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1 | 4 | 0 | 2 | 3 | 0 | 0 | 1 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 3 | 0 | 2 | 2 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 3 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Tinea capitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 2 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asymptomatic bacteriuria (Infections and infestations) | 1 | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 2 | 1 | 0 | 4 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 2 | 1 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Eschar (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood urine present (Investigations) | 0 | 2 | 0 | 2 | 4 | 2 | 2 | 1 | 5 | 2 | 2 | 2
Protein urine present (Investigations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 7 | 2 | 1 | 3 | 2 | 2 | 0 | 1 | 0 | 0 | 0
Leukocyturia (Renal and urinary disorders) | 1 | 3 | 3 | 2 | 1 | 3 | 1 | 0 | 0 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Testicular retraction (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 0 | 5 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1/16 | 0 | 0 | 0 | 0 | 0 | 0 — Number of participants at risk in the OnabotulinumtoxinA 200 U (Treatment Cycle 2) arm group is based on the female population.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-02-20): https://cdn.clinicaltrials.gov/large-docs/58/NCT01852058/SAP_000.pdf
  • Study Protocol (2016-04-14): https://cdn.clinicaltrials.gov/large-docs/58/NCT01852058/Prot_001.pdf